CLINICAL TRIAL: NCT07035184
Title: A Comparative Study Between Age-Based and Weight-Based Bupivacaine Dosing for Pediatric Spinal Anesthesia in Children Undergoing Elective Infra-Umbilical Surgeries: A Randomized Double-Blinded Controlled Trial
Brief Title: A Comparative Study Between Age-Based and Weight-Based Bupivacaine Dosing for Pediatric Spinal Anesthesia in Children Undergoing Elective Infra-Umbilical Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohammed El-Hadi Shoukat Mohammed, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: "MS-503-2024"
Record Dates: First submitted 2025-06-07; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2024-12

CONDITIONS: Pediatrics; Spinal Aneshtesia; Infraumbilical Surgeries
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: weight-based formula group (Active Comparator): Children will receive spinal anesthesia according to the weight-based dosing calculation of Hyperbaric bupivacaine 0.5% as following: 0.4 mg/kg (0.08 ml/kg) for children weighing 5-15 kg or 0.3 mg/kg (0.06 ml/kg) for children weighing >15 kg
  Interventions: Procedure: Spinal Anesthesia with Bupivacaine
- Group B: Age-based formula group (Active Comparator): Children will receive spinal anesthesia according to the age-based dosing calculation of bupivacaine. Hyperbaric bupivacaine 0.5% will be calculated using Partha formula by dividing the child's age in years by 5. The resultant figure will be considered to be the dose of Bupivacaine in ml. If the number of months after the completion of a year in age is more than 6 months, the child's age will be noted to be the year older.
  Interventions: Procedure: Spinal Anesthesia with Bupivacaine

INTERVENTIONS:
Procedure: Spinal Anesthesia with Bupivacaine — Group A (n=30) will receive spinal anesthesia according to the weight-based dosing calculation of bupivacaine.
  Arms: Group A: weight-based formula group
Procedure: Spinal Anesthesia with Bupivacaine — Group B (n=30) will receive spinal anesthesia according to the age-based dosing calculation of bupivacaine.
  Arms: Group B: Age-based formula group

SUMMARY:
This prospective randomized double-blinded controlled trial will include 60 pediatric patients aged 1 - 6 years old, both sexes, with American society of anesthesiologists (I and II) and undergoing elective infra-umbilical surgeries with anticipated duration ≤ 90 minutes. Patients will be randomly divided into two equal groups: Weight-based dosing (Group A) and age-based dosing group (Group B). Both groups will receive hyperbaric bupivacaine 0.5%. The aim of the study is to evaluate the effectiveness of using age based dosing of Bupivacaine compared with standard method of weight based dosing in pediatric spinal anesthesia.

DETAILED DESCRIPTION:
This prospective randomized double-blinded controlled trial will be conducted on 60 pediatric patients who will undergo elective infra-umbilical surgeries, e.g., inguinal hernia repair, orchiopexy, etc. admitted to the operating theatres of Abu El Reesh Children's Hospital, Cairo University.

Randomization and blinding An online randomization program (http://www.randomizer.org) will be used to generate a random list, and each patient's code will be kept in an opaque sealed envelope. Patients will be randomly allocated in a 1:1 allocation ratio into two equal groups in a parallel manner:

* Group A (n=30): Children will receive spinal anesthesia according to weight-based dosing calculation of bupivacaine
* Group B (n=30): Children will receive spinal anesthesia according to age-based dosing calculation of bupivacaine. The patient and/or related guardian will be blinded to group assignment as well as the anesthesiologist involved in data collection and analysis. A physician who is not involved in the study prepared the interventional medications.

Methods:

All patients will be subjected to the followings:

1. History taking and demographic data collection (age, sex, weight, and ASA).
2. Complete clinical examination.
3. Routine Laboratory investigations

All patients will be instructed to fast according to the following guidelines:

2 hours for clear fluids, 4 hours for breastmilk, 6 hours for formula milk and other particulate fluids. EMLA cream (5%) will be applied to the anticipated puncture sites for IV cannulation and covered for 45 minutes before transport to the OR, to facilitate the insertion of an intravenous (IV) cannula. Premedication included intramuscular (IM) midazolam at 0.3 mg/kg and atropine at 0.02 mg/kg, administered 15 minutes before transportation to the operating room (OR). Upon arrival in the OR, standard monitoring equipment will be applied, including electrocardiography, non-invasive blood pressure, and pulse oximetry. The anesthesia machine and all necessary equipment and medications for general anesthesia (GA) will be prepared for each patient. The IV cannula will be inserted, secured and checked with a saline flush. IV midazolam at a dose of 0.1 mg/kg will be given at the time of spinal anesthesia administration to ensure immobility during the procedure.

A Pediatric Analog Sedation Score (PASS) will be used to evaluate sedation levels during the procedure as well as intraoperatively, where a score of 0 = no sedation, 1 = slightly sedated, 2 = moderately sedated, 3 = well sedated, and 4 = heavily sedated. The target sedation score is 1, indicating minimal sedation. The child will be positioned in the lateral decubitus position, and under strict aseptic conditions, the lumbar region will be sterilized using Betadine. A lumbar puncture will be performed at the L4-L5 interspace (Tuffier's line) using a 2.5-inch 22-gauge Quincke needle by an experienced anesthesiologist. A formula will be used to estimate the distance from skin to subarachnoid space (mm) = [2 × weight (kg)]+ 7(mm). This will be used as a guide to reduce chances of inserting the spinal needle too deep. Two attempts at obtaining a free flow of cerebrospinal fluid (CSF) will be allowed; if unsuccessful, the patient will be excluded from the study and switched to GA. A new attempt involves removing the needle and reinserting it. The calculated dose of hyperbaric bupivacaine 0.5% (Trade name: Sunnypivacaine, Manufacturer: Sunny Pharmaceuticals, Country: Egypt) will be aspirated and administered via a 3-ml syringe.

Group A:

Hyperbaric bupivacaine 0.5% will be administered based on weight:

* 0.4 mg/kg (0.08 ml/kg) for children weighing 5-15 kg
* 0.3 mg/kg (0.06 ml/kg) for children weighing >15 kg.

Group B:

Hyperbaric bupivacaine 0.5% will be calculated using Partha formula by dividing the child's age in years by 5. The resultant figure will be considered to be the dose of Bupivacaine in ml. If the number of months after the completion of a year in age is more than 6 months, the child's age will be noted to be the year older.

After obtaining free flow of CSF, and negative aspiration test for blood, the local anesthetic will be administered slowly. Then, the child will be placed in a supine position with a small pillow under the head. IV fluids will be administered at a rate of 4 ml/kg/hr. Sensory and motor levels will be assessed every minute for the first 5 minutes. The adequacy of the block will be determined by the lack of response to a firm skin pinch at the dermatomal level. The peak sensory level will be determined when the dermatomal level remained unchanged in at least two consecutive assessments. If the patient reported pain, the block will be considered failed, and they are excluded from the study. Motor blockade at or above the L1 level will be tested using superficial abdominal reflexes. After a maximum of ten minutes after spinal anesthesia, the target peak sensory level should be at least T10, and the Bromage score should be 3, indicating a complete motor block. Only then the surgery will be proceeded. Iff inadequate sensory or motor block are observed (e.g., peak sensory level below T10 or Bromage score <3), GA will be administered, and the failure will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-6 years

  * Both genders.
  * American Society of Anesthesiologists (ASA) physical status I or II.
  * Elective infra-umbilical surgeries with anticipated duration ≤ 90 minutes.

Exclusion Criteria:

* Guardian refusal.

  * Children with significant congenital heart disease (e.g., septal defects requiring surgical intervention)
  * Children with neuromuscular disorders or high intracranial pressure.
  * Children with spinal deformities or morbid obesity (body mass index (BMI) above the 99th percentile).
  * Children with a history or family history of coagulation disorders.
  * Children with local infection at the site of skin puncture for spinal anesthesia.
  * Children with known allergy to Bupivacaine.
  * Surgeries requiring Trendelenburg or prone position.
  * Unexpected prolongation of surgery > 90 minutes

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
The peak sensory level | Assessed 5 minutes after intrathecal bupivacaine injection, and evaluated by a firm skin pinch up to 30 minutes after subarachnoid block
  The peak sensory level will be assessed 5 minutes after intrathecal bupivacaine injection, and evaluated by a firm skin pinch.

SECONDARY OUTCOMES:
Time of completion of spinal block | starts immediately at the time of application of Betadine on the site of lumbar puncture to the time at which the patient is placed on their back after immediately administering the spinal anesthesia
  Time in seconds to complete block administration starting at the time of application of Betadine on the site of lumbar puncture to the time at which the patient is placed on their back after administration of spinal anesthesia
Duration of spinal block | starts immediately after achieving a peak sensory and motor levels and eds immediately by the onset of perioperative pain or movement of legs
  Duration of block: the time in minutes from achieving peak sensory and motor level to the onset of pain or the movement of the legs.
Postoperative pain score | Scale will be assessed postoperatively at 2 hours, 4 hours, and 6 hours from block administration.
  Postoperative pain score will be recorded using the Face, Legs, Activity, Cry, and Consolability (FLACC) Scale at 2, 4, and 6 hours from block administration. The scale consists of five categories: Face, Legs, Activity, Cry, and Consolability, each of which is scored from 0 to 2. A score of 0 represents no pain or distress, while a score of 2 indicates significant discomfort or distress.
The need for rescue analgesia in PACU | Postoperatively at 2 hours after spinal block and up to 1 hour postoperatively
  The need for rescue analgesia in PACU: IV Pethidine 1 mg/kg will be administered once for a pain score of 6 or higher using FLACC scale
Incidence of failure of spinal block | 20 minutes after local anesthetic administration until 30 minutes after local anesthetic administration
  Incidence of failure of spinal block defined by a failure to reach sensory level of T10 and modified Bromage score of 3; therefore, requiring the switch to GA.
Complications related to anesthesia | started immediately after lumbar puncture and followed up for 2 hours postoperatively
  Complications related to anesthesia, such as vomiting, shivering, post dural puncture headache, and any manifestation suggestive of neurological injury, will be recorded.
Incidence of intraoperative complications | Started immediately after spinal block until the end of surgery
  Incidence of hypotension and or bradycardia defined as and 20% decrease from baseline values

OTHER OUTCOMES:
Systolic blood pressure (SBP) | Will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery until the end of surgery.
  SBP will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery.
Diastolic blood pressure (DBP) | Will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery until the end of surgery.
  DBP will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery.
Mean blood pressure (MBP) | Will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery until the end of surgery.
  MBP will be recorded at T0 (baseline values before administration of block), then upon administration of spinal anesthesia, then every 3 minutes for 15 minutes, then every 5 minutes for the duration of the surgery.
The dose bupivacaine administered. | Before the administration of local anesthesia, the dose will be calculated according to the group until the preoperative administration of spinal block.
  The dose in millilitres of bupivacaine administered in each group will be recorded.
Duration of surgery | Perioperatively
  duration of surgery in minutes
Type of surgery | Perioperatively
  type of infraumbilical surgery
Age of patients | Perioperatively
  Age in years will be recorded
Sex of patients | Recorded immediately preoperatively until immediately before lumbar puncture
  Patients' gender
Weight of patients | Started immediately preoperatively until immediately before lumbar puncture
  Weight in Kilograms will be recorded
ASA status | Started immediately preoperatively until immediately before lumbar puncture
  American Society of Anesthesia physical status (ASA), ranged from I to IV. Only I & II included in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Abu Elreesh Pediatric Hospital, Cairo, Assida Zainab, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publications

REFERENCES:
- [Background] Crellin DJ, Harrison D, Santamaria N, Huque H, Babl FE. The Psychometric Properties of the FLACC Scale Used to Assess Procedural Pain. J Pain. 2018 Aug;19(8):862-872. doi: 10.1016/j.jpain.2018.02.013. Epub 2018 Mar 15. PMID 29551662
- [Background] Srinivasan P, Saravanan B, Kulandayan I, Thambidurai S, Mahalakshmi V. Evaluation of efficacy and safety of age-based intrathecal dosing of 0.5% hyperbaric bupivacaine in the paediatric age group. J Clin Diagn Res. 2020;14(8):29-31.
- [Background] Troncin R, Dadure C. Paediatric spinal anaesthesia. management. 2009;4(3):8-12.
- [Background] Elsharkawi NG. Simple pediatric analog sedation score (PASS). Anesth Analg. 1999 Jan;88(1):227. doi: 10.1097/00000539-199901000-00043. No abstract available. PMID 9895098
- [Background] Luca E, Schipa C, Cambise C, Sollazzi L, Aceto P. Implication of age-related changes on anesthesia management. Saudi J Anaesth. 2023 Oct-Dec;17(4):474-481. doi: 10.4103/sja.sja_579_23. Epub 2023 Aug 18. PMID 37779561
- [Background] Hebbes CP, Thompson JP. Pharmacokinetics of anaesthetic drugs at extremes of body weight. BJA Educ. 2018 Dec;18(12):364-370. doi: 10.1016/j.bjae.2018.09.001. Epub 2018 Oct 26. No abstract available. PMID 33456803
- [Background] Visavakul O, Leurcharusmee P, Pipanmekaporn T, Khorana J, Patumanond J, Phinyo P. Effective Dose Range of Intrathecal Isobaric Bupivacaine to Achieve T5-T10 Sensory Block Heights for Elderly and Overweight Patients: An Observational Study. Medicina (Kaunas). 2023 Mar 1;59(3):484. doi: 10.3390/medicina59030484. PMID 36984485
- [Background] Parthasarathy S, Senthilkumar T. Age-based Local Anesthetic Dosing in Pediatric Spinal Anesthesia: Evaluation of a New Formula - A Pilot Study in Indian Patients. Anesth Essays Res. 2017 Jul-Sep;11(3):627-629. doi: 10.4103/aer.AER_246_16. PMID 28928560
- [Background] Lonnqvist PA. Spinal anaesthesia in children: A narrative review. Best Pract Res Clin Anaesthesiol. 2023 Jun;37(2):133-138. doi: 10.1016/j.bpa.2023.01.002. Epub 2023 Feb 7. PMID 37321762
- [Background] Jefferson FA, Findlay BL, Handlogten KS, Gargollo PC, Warner LL, Woodbury JM, Haile DT, Granberg CF. Spinal anesthesia in infants undergoing urologic surgery duration greater than 60 minutes. J Pediatr Urol. 2022 Dec;18(6):786.e1-786.e7. doi: 10.1016/j.jpurol.2022.07.003. Epub 2022 Jul 14. PMID 35945145
- [Background] Verma D, Naithani U, Gokula C, Harsha. Spinal anesthesia in infants and children: A one year prospective audit. Anesth Essays Res. 2014 Sep-Dec;8(3):324-9. doi: 10.4103/0259-1162.143124. PMID 25886329
- [Background] Heydinger G, Tobias J, Veneziano G. Fundamentals and innovations in regional anaesthesia for infants and children. Anaesthesia. 2021 Jan;76 Suppl 1:74-88. doi: 10.1111/anae.15283. PMID 33426659